CLINICAL TRIAL: NCT05246592
Title: Postoperative Upper Limb Edema and Dysfunction Generated by Axillary Nodes Excision Differs Due to the Ratio of Axillary Lymphatic and Axillary Vein Reflux in Breast Cancer Patients: a Prospective Cohort Study
Brief Title: Effect of the Axillary Lymphatic /Vein Reflux Ratio on Postoperative Upper Limb Edema and Dysfunction in Breast Cancer
Acronym: PLEDGE-R
Status: Active, not recruiting | Type: Observational
Sponsor: Xiangyun Zong (Other)
Responsible Party: Sponsor-Investigator, Xiangyun Zong, Head of Breast Cancer, Principal Investigator, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Other Study IDs: JTU-6H-20211230001
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Lymphedema
Keywords: Breast Cancer; Axillary Lymph Node Dissection; Post-mastectomy Lymphedema; Upper Limb Dysfunction; axillary lymphatic reflux; axillary vein reflux
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preponderant lymphatic reflux group: high ratio of axillary lymphatic reflux to axillary vein reflux
  Interventions: Procedure: Branches Sparing; Procedure: None Branches Sparing
- Preponderant venous reflux group: low ratio of axillary lymphatic reflux to axillary vein reflux
  Interventions: Procedure: Branches Sparing; Procedure: None Branches Sparing

INTERVENTIONS:
Procedure: Branches Sparing — The patients will undergo axillary lymph node dissection with preserved axillary vein branches
Procedure: None Branches Sparing — The patients will undergo axillary lymph node dissection without preserved axillary vein branches

SUMMARY:
The purpose of this study is to compare the difference in the incidence of upper limb edema and dysfunction between the Preponderant lymphatic reflux group (high ratio of axillary lymphatic reflux to axillary vein reflux) and the Preponderant venous reflux group (low ratio of axillary lymphatic reflux to axillary vein reflux).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years old,
* Regardless of gender,
* Breast masses were diagnosed by histology and pathology, stage II -III.
* Clinical palpation of axillary lymph nodes is positive, or
* Axillary lymph node puncture pathology is positive, or
* The multidisciplinary treatment cooperation group (MDT) recommends axillary lymph node dissection,
* Good physical state score (0-1),
* No severe organ complications,
* No congenital or acquired diseases affecting the normal morphology and functional activities of the upper limbs,
* Informed consent, understanding and compliance with research requirements.

Exclusion Criteria:

* Pregnancy or lactation,
* Inflammatory breast cancer,
* Clinical findings of metastatic lesions,
* Sentinel lymph node biopsy was negative,
* History of upper limb or shoulder, chest, back trauma or surgery,
* Previous history of local radiotherapy,
* History of other tumors,
* Vascular embolic disease,
* Those who are unable to comply with the clinical trial requirements for any reason.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited in the PLEDGE study （NCT05120180）
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
short-term Incidence of lymphedema | 1-, 6-, and 12-month
  Incidence of upper limb lymphedema on affected side at 1-, 6-, and 12-month after operation
short-term Incidence of dysfunction | 1-, 6-, and 12-month
  Incidence of upper limb dysfunction on affected side at 1-, 6-, and 12-month after operation

SECONDARY OUTCOMES:
long-term Incidence of lymphedema | 5 years
  Incidence of upper limb lymphedema on affected side 5 years after operation
long-term Incidence of dysfunction | 5 years
  Incidence of upper limb dysfunction on affected side 5 years after operation

OTHER OUTCOMES:
Risk model | 5 years
  To establish a risk model of upper limb edema and dysfunction after axillary dissection for breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: XIANGYUN ZONG, MD, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shanghai Fengxian Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No